CLINICAL TRIAL: NCT06306651
Title: Comparative Study Between High Flow Nasal Cannula and Conventional Oxygen Therapy in the Postoperative Management of Patients With Mild to Moderate Obstructive Sleep Apnea
Brief Title: High Flow Nasal Cannula and Conventional Oxygen Therapy in the Postoperative Management of Patients With Mild to Moderate Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar medhat, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD283/2023
Record Dates: First submitted 2024-03-03; First posted 2024-03-12 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: High Flow Nasal Cannula; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High flow nasal cannula therapy group (Experimental): Patients who will be randomized to high flow nasal cannula therapy. High flow nasal oxygen cannula will be applied at a flow of 20 L/min at FiO2 of 0.4 at a temperature of 36oC.
  Interventions: Other: High flow nasal cannula therapy group
- Conventional oxygen therapy group (Active Comparator): Patients who will be randomized to simple oxygen mask therapy. The simple face mask will be applied in a rate range between 6-10 L/min.
  Interventions: Other: Conventional oxygen therapy group

INTERVENTIONS:
Other: High flow nasal cannula therapy group — Patients who will be randomized to high flow nasal cannula therapy. High flow nasal oxygen cannula will be applied at a flow of 20 L/min at FiO2 of 0.4 at a temperature of 36oC
  Arms: High flow nasal cannula therapy group
Other: Conventional oxygen therapy group — Patients who will be randomized to simple oxygen mask therapy. The simple face mask will be applied in a rate range between 6-10 L/min.
  Arms: Conventional oxygen therapy group

SUMMARY:
This study aims to compare the effectiveness of conventional oxygen therapy oxygen and high-flow nasal cannula therapy on oxygen saturation (SpO2), measuring number of SpO2 drop >4% of base line oxygen saturation (o2 desaturation index), length of the ICU stay, and the need of use supplemental continuous positive airway pressure (CPAP) support in any of the study groups in the postoperative ICU setting.

DETAILED DESCRIPTION:
In the surgical setting, patients with obstructive sleep apnea (OSA) may have increased upper airway collapsibility affecting ventilation and increased sensitivity to sedation from anesthetics and opioids.

Surgical patients with OSA have a high risk for postoperative complications, including cardiac events, hypoxemia, and transfer to the intensive care unit . Continuous positive airway pressure (CPAP) is the gold standard treatment for moderate to severe OSA , and effectively reduces the risk of cardiovascular events. Evidence has shown that CPAP effectively reduces length of ICU stay (LOS) in the postoperative setting. In these scenarios, conventional oxygen therapy and high-flow nasal cannula (HFNC) therapy have been used as an alternative for CPAP non-adherent patients.

HFNC delivers warm, humidified air through a nasal cannula at high flow rates of up to 60 L/min. This high flow rate may increase end-expiratory pharyngeal pressure up to 3 cm H2O, decreasing the force required to alleviate airway collapse . Using a nasal cannula interface in contrast to the CPAP mask may provide a more comfortable experience for patients during sleep .

ELIGIBILITY:
Inclusion Criteria:

* Age group from 21 - 40 years old.
* Both sexes.
* Mild to moderate obstructive sleep apnea (OSA) patients with STOP-BANG score less than 5.
* OSA patients undergoing non cardiac surgeries.
* Patients who will undergo scheduled elective surgeries under general anesthesia.

Exclusion Criteria:

* Patient refusal of procedure or participation in the study.
* Patients with severe OSA, STOP-BANG score more than or equal 5.
* Patients dependent on home ventilation CPAP or bilevel devices.
* Pregnant females.
* Post cardiac or thoracic surgery patients.
* More than American Society of Anesthesiologists (ASA) II patients.
* Head and face trauma patients.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen desaturation index | During intensive care unit stay (assessed up to day 5)
  Oxygen desaturation index will be recorded through by pulse oximeter, while respiratory rate will be recorded by the ECG monitoring and visual count hourly.
  The number of recorded drops in baseline SpO2 of >4%.

SECONDARY OUTCOMES:
The length of Intensive care unit stay | At the time of intensive care unit discharge (up to day 5)
  The length of Intensive care unit stay will be measured from the start of surgery until the discharge.
The incidence of ventilatory support | At the time of intensive care unit discharge (up to day 5)
  The incidence of ventilatory support is either non-invasive ventilation (NIV) and continuous positive airway pressure (CPAP) or intubation and mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.